CLINICAL TRIAL: NCT02665936
Title: Epidural Levobupivacaine Versus A Combination of Levobupivacaine and Dexamethasone in Parturients Receiving Epidural for Vaginal Delivery Analgesia: A Comparative, Dose Ranging and Safety Evaluation Study
Brief Title: Effect of Epidural Dexamethasone on Labor Analgesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, ahmed elsakka, m.d. anasthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: wahdan
Record Dates: First submitted 2016-01-13; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Labor
Keywords: epidural analgesia
MeSH Terms: interventions — Levobupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- group L (Active Comparator): Epidural levobupivacaine 0.125% (Chirocaine) in normal saline in a total volume of 10 ml will be administered epidurally in active stage of labor
  Interventions: Drug: Levobupivacaine
- group LD4 (Active Comparator): Epidural levobupivacaine 0.125%(Chirocaine) in normal saline combined with dexamethasone 4 mg in a total volume 10 ml
  Interventions: Drug: Dexamethasone and levobupivacaine
- group LD8 (Active Comparator): Epidural levobupivacaine 0.125%(Chirocaine) in normal saline combined with dexamethasone 8 mg in a total volume 10 ml
  Interventions: Drug: Levobupivacaine and Dexamethasone

INTERVENTIONS:
Drug: Levobupivacaine — Levobupivacaine will be given epidurally and the duration of analgesia will be calculated
  Arms: group L
Drug: Dexamethasone and levobupivacaine — dexamethasone 4 mg epidurally with levobupivacaine and duration of analgesia is measured
  Arms: group LD4
Drug: Levobupivacaine and Dexamethasone — dexamethasone 8 mg epidurally with levobupivacaine and duration of analgesia is measured
  Arms: group LD8

SUMMARY:
The purpose of this study is to detect whether the addition of epidural dexamethasone will prolong labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II
* normal vaginal delivery In early active phase of labor
* singleton cephalic presentation at term

Exclusion Criteria:

* complicated pregnancies
* morbid obesity
* diagnosed fetal abnormalities
* contra-indications to regional anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Duration of epidural analgesia | an average of 5 months

SECONDARY OUTCOMES:
Time of onset of sensory block at level T10 | an average of 5 months
  From the onset of active stage till the end of labor

CONTACTS AND LOCATIONS:
Overall Officials: ahmed i elsakka, m,d,, Principal Investigator — Cairo University; amira r hassan, m,d., Study Chair — Cairo University; nadia y helmy, m.d., Study Director — Cairo University